CLINICAL TRIAL: NCT05338190
Title: A Phase 3 Randomized and Double-blind Controlled Trial Comparing the Efficacy and Safety of Subcutaneous Belimumab or Placebo in Addition to Rituximab in Adult Patients With Persistent or Chronic Immune Thrombocytopenia (ITP)
Brief Title: Efficacy and Safety of Subcutaneous Belimumab or Placebo in Addition of Rituximab in Persistent or Chronic Immune Thrombocytopenia
Acronym: RITUX-PLUS 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP201098; 2021-000006-16 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-04-21 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): Belimumab 200 mg subcutaneous weekly (i.e., every 7 days ±1 day) starting from day 0 through week 24 with 1 g intravenous of Rituximab 7 days and 21 days after the randomization.
  Interventions: Drug: Combination of Rituximab with subcutaneous belimumab
- ARM B (Placebo Comparator): Placebo subcutaneous weekly (i.e., every 7 days ±1 day starting from day 0) starting from day 0 through week 24 with 1 g intravenous of Rituximab 7 days and 21 days after the randomization.
  Interventions: Drug: Combination of Rituximab with subcutaneous placebo

INTERVENTIONS:
Drug: Combination of Rituximab with subcutaneous belimumab — Belimumab 200 mg subcutaneous weekly (i.e., every 7 days ±1 day) starting from day 0 through week 24 with 1 g intravenous of Rituximab 7 days and 21 days after the randomization.
  Arms: ARM A
Drug: Combination of Rituximab with subcutaneous placebo — Placebo subcutaneous weekly (i.e., every 7 days ±1 day starting from day 0) starting from day 0 through week 24 with 1 g intravenous of Rituximab 7 days and 21 days after the randomization.
  Arms: ARM B

SUMMARY:
Primary immune thrombocytopenia (ITP) is an autoimmune disease mainly mediated by autoreactive B cells and the presence of pathogenic anti-platelet auto-antibodies that enhance platelet destruction and impair platelet production. There are approximately 4,000 newly diagnosed ITP cases each year in France. For patients with a platelet count of less than 30x109/L and/or bleeding symptoms, corticosteroids alone or in combination with intravenous immunoglobulin (IVIg) is the standard first-line treatment. However, approximately two-thirds of adult patients responding to this first-line treatment relapse within days or weeks after corticosteroids withdrawal and overall, the course of the disease is chronic in about 70% of the cases. The anti-CD20 monoclonal antibody rituximab is commonly used off-label as a second-line therapy in many European countries including France for adults with persistent (i.e., disease duration of more than 3 months) or chronic (disease duration of more than 12 months) ITP. Rituximab leads to an overall response rate of only 40 % at 1 year but 29.5% of lasting (5 years and more) response The investigators have shown that the absence of response to rituximab in ITP could be explained by the settlement and expansion of long-lived autoreactive plasma cells in the spleen made possible by the high amount of BAFF. Belimumab is a fully humanized anti-BAFF/Blys monoclonal Ab licensed for SLE. Based on the preliminary results of a phase 2 open prospective pilot study performed in our center combining rituximab with i.v belimumab seems highly promising We hypothesized that combining subcutaneous belimumab weekly over a 24 weeks period (Arm A) with rituximab is superior to rituximab and subcutaneous placebo weekly over 24 weeks period (Arm B) to achieve an overall response at W52.

The study design will be a prospective randomized, double-blind, multicenter (international), superiority phase III clinical study

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Primary ITP defined according to the standard definition criteria (Rodeghiero, Blood 2008)
3. Previous response to corticosteroids and/or IgIV defined by a rise of platelet levels > 30 x 109/L with at least a twofold increase from baseline levels followed by a relapse.
4. Platelet count ≤ 30 x 109/L within the previous month or <50 x 109/L if presence of haemorrhagic events or other reason left up to investigator discretion.
5. ITP duration of more than 2 months but less than 5 years from diagnosis.
6. Normal bone marrow smear for patients above 60 years of age
7. Negative pregnancy test results and effective contraception for women of childbearing age Female subjects of childbearing potential must not become pregnant and so must be sexually inactive by abstinence or use contraceptive methods with a failure rate of < 1%.

   Therefore, these women must have a negative serum pregnancy test at screening, and confirmed monthly while in study (with serum or Urine test), out to at least 12 months (taking account of the longest half-life which is that of 29.7 days and according to smPC) post last dose and agree to 1 of the following:
   * Complete abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent until 16 weeks after the last dose of study agent (Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception) OR
   * Consistent and correct use of 1 of the following acceptable methods of birth control for 1 month prior to the start of the study agent, during the study, and 16 weeks after the last dose of study agent

     * Oral contraceptive, either combined or progestogen alone
     * Injectable progestogen
     * Implants of levonorgestrel or etonogestrel
     * Estrogenic vaginal ring
     * Percutaneous contraceptive patches
     * Intrauterine device (IUD) or intrauterine system (IUS) with <1% failure rate as stated in the product label
     * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records
     * Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring subjects understand how to properly use these methods of contraception.
8. Complete Vaccinal scheme against SARS-CoV2 according to the recommendations of the health authorities
9. Gammaglobulin level ≥ 7 g/L
10. Informed consent
11. Affiliated to, or beneficiary of, a social security regime or similar

Exclusion Criteria:

1. Splenectomy
2. Previous treatment with rituximab or any B-cell targeted therapy
3. Common variable immunodeficiency
4. Previous treatment with cyclophosphamide or ciclosporin
5. Inclusion in another clinical trial less than 3 months before inclusion
6. Previous anaphylactic shock to previous biologic therapy
7. Chronic or ongoing severe infection requiring treatment or hospitalization in the 60 days preceding inclusion.
8. Use of parenteral antibiotics within 60 days, current use of suppressive therapy for chronic infection such as tuberculosis, pneumocystis, cytomegalovirus, HSZ, herpes zoster, and atypical mycobacteria
9. Evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.
10. Psychiatric Illness impairing judgement.
11. Neutrophils count < 1,000/mm3 at inclusion
12. Positive HIV test and/or hepatitis virus C infection and/or positive hepatitis B virus surface antigen or core antibody (HbsAg or HBcAb)
13. Impaired renal function as indicated by a serum creatinine level > 2 mg/dl
14. Liver function: AST (SGOT) and ALT (SGPT) ≥5xULN Total bilirubin ≥3 x ULN
15. New York Heart Classification III or IV heart disease
16. Previous history of malignancy in the last 5 years other than cutaneous carcinoma
17. Previous history of Progressive multifocal leukoencephalopathy
18. Previous history of major organ transplant or hematopoietic stem cell/marrow transplant or renal transplant.
19. Alcohol or drug abuse or dependence, either current or within 1year
20. Pregnant or breast-feeding woman
21. Live, attenuated vaccinations must be administered at least 30 days before inclusion in study
22. History of significant medical illness or clinically significant laboratory abnormality (or planned surgical procedure) which in the opinion of the investigator would interfere with the study procedures and / or assessments or compromise subject safety
23. Body mass index > 40
24. PCR-confirmed SARS-CoV-2 infection
25. Vulnerable persons, under the protection of justice,
26. Persons deprived of their liberty by judicial or administrative decision,
27. Persons admitted to a health or social establishment for purposes other than research,
28. Persons under legal protection (guardianship, curatorship),
29. Persons unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-11-14 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (CR + R) in both arms at W52 | Week 52
  To assess the superiority at W52 of a combination subcutaneous belimumab weekly over a 24 weeks period (Arm A) or subcutaneous placebo weekly during 24 weeks period (Arm B) with rituximab (or biosimilar) (at a fixed dose of 1,000 mg on Day 7 and Days 21).

SECONDARY OUTCOMES:
Number of patients developing a severe hypogammaglobulinemia in both arms | at Week 12, Week 24, Week 36, Week 52, Week 88, Week 104
  (gammaglobulin level < 4 g/dl)
Duration of a severe hypogammaglobulinemia | up to Week 104
  Duration of a severe hypogammaglobulinemia in patients with such complication
Variation in gammaglobulin | Frame throughout the study (Week 0, Week 12, Week 24, Week 36, Week 52, Week 88, Week 104)
  Variation in gammaglobulin classes and subclass levels
Number of severe infections | up to Week 104
  Number of severe infections requiring hospitalization
Platelet levels | at Week 6, Week 12, Week 24, Week 36, Week 52, Week 88, Week 104
Total number of responders | at Week 6, Week 12, Week 24, Week 36, Week 52, Week 88, Week 104
Number of haemorrhagic events | at Week 6, Week 12, Week 24, Week 36, Week 52, Week 88, Week 104.
Percentage of each B-cell subpopulation, T Follicular helper population and levels of cytokines including BAFF and anti-platelet antibodies | at Week 12, Week 24, Week 36, Week 52, Week 88, Week 104

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, France